CLINICAL TRIAL: NCT06600815
Title: Analgesic Efficacy of Preemptive Stepwise Infiltration Anesthesia for Perioperative Analgesia After Total Knee Arthroplasty: a Prospective Double-blind Randomized Controlled Clinical Trial
Brief Title: Analgesic Efficacy of Preemptive Stepwise Infiltration Anesthesia for Perioperative Analgesia After TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Fang, Deputy chief physician, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRCTA, ECFAH of FMU|2024]576
Record Dates: First submitted 2024-08-02; First posted 2024-09-19 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Total Knee Arthroplasty; Pain Management
Keywords: Total knee arthroplasty; Pain management; Anaesthesia in orthopaedics
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The trial employs a random allocation method. A randomization table will be generated using SPSS 26.0 software. Treatment groups will be selected based on patients' random numbers, ensuring that this clinical institution stratifies the subjects into a PSIA group and a PLIA group at a 1:1 ratio.
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers, outcome assessors and statisticians will be blinded to the group assignments and will not be involved in the trial operations. The patients will also be blinded to the group assignments. Due to the impossibility of blinding the surgeons, they will not be involved in any outcome assessments. Allocation results will be placed in sealed envelopes before the surgery. The envelopes will be opened prior to surgery after the administration of general anaesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- preemptive stepwise infiltration anaesthesia(PSIA) group (Experimental): Drugs：A cocktail of anaesthetics (30 mg of ropivacaine, 0.3 mg of adrenaline) will be prepared, diluted with normal saline to 120 mL, and divided into two equal parts(Cocktail A[CA] and Cocktail B[CB]), with CB containing 8 mg of added betamethasone (each 1 ml of the compound contains 5 mg betamethasone dipropionate [calculated as betamethasone] and 2 mg of betamethasone sodium phosphate [calculated as betamethasone]).
  Interventions: Procedure: preemptive stepwise infiltration anaesthesia(PSIA)
- postoperative local infiltration analgesia(PLIA) group (Active Comparator): Drugs: the same preoperative preparation and treatment with the anaesthesia cocktail formulation as those in the PSIA group.
  Interventions: Procedure: postoperative local infiltration analgesia(PLIA)

INTERVENTIONS:
Procedure: preemptive stepwise infiltration anaesthesia(PSIA) — For PSIA patients, the anaesthetic is administered in stages. Initially, CA is injected at the incision site before the medial parapatellar incision. Following skin incision, more CA is injected into the subcutaneous tissue. After exposing the fascial layer and joint capsule, CA is used around the patellar tendon, and then CB is injected into the joint capsule and surrounding muscles. Additional CB is applied to the synovium and soft tissues after the joint cavity is opened, and more is used in the posterior joint capsule after bone resection.
  Arms: preemptive stepwise infiltration anaesthesia(PSIA) group
Procedure: postoperative local infiltration analgesia(PLIA) — Before standardized TKA and implantation of the prosthesis, 30-40 mL of CB will be used to infiltrate the synovium and whole joint capsule. Subsequently, the joint cavity, subcutaneous tissue, and skin will be closed layer by layer using routine procedures. After the skin is closed, 30-40 mL of CA will be injected into the skin and subcutaneous tissue.
  Arms: postoperative local infiltration analgesia(PLIA) group

SUMMARY:
This is a single-center prospective cohort study in which patients were evaluated by inclusion and exclusion criteria before total knee arthroplasty (TKA). Eligible patients will be included in this study after signing the informed consent form. Before TKA, the patients will be randomly assigned to either a preemptive stepwise infiltration anaesthesia (PSIA) group or a postoperative local infiltration analgesia (PLIA) group and administered different pain management protocols during surgery. Clinical evaluation will be conducted at baseline, before surgery, and at 6, 12, 24, 48, and 72 hours postoperatively, as well as during follow-up visits at 3 weeks, 6 weeks and 6 months postoperatively. All patients voluntarily participated in the study and signed informed consent. During the treatment period, all prospective patients underwent clinical evaluation at the end of total knee arthroplasty and 6, 12, 24, 48, 72, and 96 weeks later, aimed at comparing the postoperative pain and inflammatory response between PSIA and PLIA, to explore the optimal perioperative analgesic modality for TKA.

DETAILED DESCRIPTION:
This is a single-center prospective cohort study in which patients were evaluated by inclusion and exclusion criteria before total knee arthroplasty (TKA). This study aims to recruit 110 patients across a single centre over 1 year. Eligible patients will be included in this study after signing the informed consent form. Before TKA, the patients will be randomly assigned to either a preemptive stepwise infiltration anaesthesia (PSIA) group or a postoperative local infiltration analgesia (PLIA) group and administered different pain management protocols during surgery. Clinical evaluation will be conducted at baseline, before surgery, and at 6, 12, 24, 48, and 72 hours postoperatively, as well as during follow-up visits at 3 weeks, 6 weeks and 6 months postoperatively. The primary outcomes are the amount of morphine consumed within 0-24 hours postsurgery and the visual analogue scale (VAS) score postsurgery. Secondary outcomes include the time to first rescue analgesia, total morphine consumption during hospitalization, postoperative joint function (measured by the Hospital for Special Surgery [HSS] score and knee joint range of motion [ROM]), intraoperative bleeding and serological indicators. All patients voluntarily participated in the study and signed informed consent. During the treatment period, all prospective patients underwent clinical evaluation at the end of total knee arthroplasty and 6h, 12h, 24h, 48h, 72h, 3 weeks, 6 weeks and 6 months later, aimed at comparing the postoperative pain and inflammatory response between PSIA and PLIA, to explore the optimal perioperative analgesic modality for TKA. Statistical analyses utilizing regression models and survival analysis will be conducted to assess the relationships between the pain management method and postoperative pain and efficacy.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for inclusion:

1. Clinical diagnosis of primary unilateral knee osteoarthritis (KOA), confirmed by imaging as KOA (Kellgren-Lawrence score ≥2). The patient was scheduled for initial unilateral total knee arthroplasty (TKA) at our hospital.
2. Preoperative American Society of Anaesthesiologists (ASA) score ranging from 1 to 3. Surgeons deemed the patient eligible for TKA based on the evaluation criteria.
3. Participants aged 18 years or older, both male and female.
4. Ability to provide informed consent and sign a written informed consent form.
5. The ability to comprehend the research requirements and willingness to cooperate with the study instructions.

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

1. Previous knee surgery on the operative knee or a history of infection in the operative knee.
2. Patients diagnosed with conditions other than osteoarthritis (including rheumatoid arthritis, traumatic arthritis, septic arthritis and haemophilic arthritis).
3. Severe osteoarthritis (including flexion contracture >30° or varus/valgus deformity >30° and the use of unconventional arthroplasty components due to complex joint pathology [e.g., restrictive prostheses]).
4. Allergy to the investigational drug.
5. The presence of neuromuscular dysfunction on the operative side.
6. Dependence on anaesthesia drugs (defined as the use of opioid or local anaesthetic drugs exceeding 100 mg of morphine equivalents per week to control preoperative pain for more than 3 months).
7. Poor overall health conditions, including but not limited to a glycated haemoglobin level exceeding 12%; blood pressure exceeding 170/110 mmHg; myocardial infarction, stroke, transient ischaemic attack, acute congestive heart failure, or any acute coronary events within the past 6 months; severe hepatic or renal dysfunction; and pregnancy or lactation.
8. Concurrent participation in clinical trials other than this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine consumption within the first 24 hours | the first 24 hours after TKA
  Postoperative morphine consumption within the first 24 hours includes both routine analgesia and rescue analgesia, which will be converted to oral morphine equivalents (OMEs)
. Postoperative visual analogue scale (VAS) scores at 6 hours, 12 hours, 24 hours, 48 hours, 72 hours, 3 weeks, 6 weeks and 6 months | 6 hours, 12 hours, 24 hours, 48 hours, 72 hours, 3 weeks, 6 weeks and 6 months after TKA
  VAS scores are the most commonly used indicator for assessing the intensity of patient pain (15). The scale ranges from "0" to "10", where "0" indicates no pain and "10" represents the most severe pain that is unbearable. Patients will rate their pain based on subjective perceptions. In this trial, VAS scores will be recorded once before TKA. The VAS scores will be assessed separately for the resting and flexion states. If the patient's hospitalization period is shorter than 72 hours, the VAS score at discharge will be recorded instead of that at 72 hours. Studies have shown that some patients still experience joint pain six months after TKA. The VAS scores of patients at 6 months after TKA will be evaluated. A VAS score of 4 or above is defined as "chronic persistent pain after TKA." The results will be used to evaluate whether PSIA can reduce pain after TKA.

SECONDARY OUTCOMES:
Postoperative time to first rescue analgesia | up to 3 days
  Rescue analgesia will be initiated when the patient reports local knee joint pain on the operative side with a VAS score > 4. The specific steps will be implemented as described previously. The time to rescue analgesia will be recorded.
Total morphine consumption during hospitalization | through study completion, an average of 6 months
  It will be converted to total morphine equivalents and will include both the postoperative routine pain management regimen and rescue analgesia.
The Hospital for Special Surgery Knee Score (HSS) | 3 weeks, 6 weeks and 6 months postoperatively
  The Hospital for Special Surgery Knee Score (HSS) is a patient-reported questionnaire specific to the knee joint, with a total score of 100 points. It comprises six scoring components: pain (30 points), function (22 points), range of motion (18 points), muscle strength (10 points), knee deformity (10 points) and stability (10 points). Additional points are deducted for the use of assistive devices, extension lag and varus deformity: up to 3 points for assistive device use, up to 5 points for extension lag and 1 point deducted for every 5 degrees of varus deformity. The scores are classified as follows: ≥ 85 as "Excellent", 70-84 as "Good", 60-69 as "Fair", and < 60 as "Poor". The HSS score is widely praised for its perceived ease of use and quick recording and has been shown to be an effective and reliable measure for assessing the efficacy of TKA.
Range of motion (ROM) | 3 weeks, 6 weeks and 6 months postoperatively
  The range of motion (ROM) will be measured with a protractor thrice daily at 6-hour intervals, and the best value on each day will be used in the analysis. The range of motion (ROM) is from 0 to 180 degrees. The larger the angle, the more satisfactory the recovery of joint function.
Direct intraoperative bleeding | 24 hours postoperatively
  Intraoperative bleeding will be recorded directly by anesthesiologists (mL).
Indirect intraoperative bleeding | 24 hours postoperatively
  Intraoperative bleeding will be estimated by subtracting the preoperative hemoglobin level from the hemoglobin level measured 24 hours postoperatively.
Complete blood count | 72 hours, 3 weeks, 6 weeks and 6 months postoperatively
  A complete blood count (CBC) can reflect the patient's postoperative inflammatory status. It measures various components of the blood, including white blood cells, red blood cells, and platelets, which can indicate the presence of inflammation or infection. An elevated white blood cell count, for example, is often associated with an inflammatory response.
C-reactive protein (CRP) | 72 hours, 3 weeks, 6 weeks and 6 months postoperatively
  C-reactive protein (CRP) can reflect the patient's postoperative inflammatory status.
Erythrocyte sedimentation rate (ESR) | 72 hours, 3 weeks, 6 weeks and 6 months postoperatively
  Erythrocyte sedimentation rate (ESR) can reflect the patient's postoperative inflammatory status.
Interleukin-6 (IL-6) | 72 hours, 3 weeks, 6 weeks and 6 months postoperatively
  Interleukin-6 (IL-6) can reflect the patient's postoperative inflammatory status.
Total bilirubin (TB) | 72 hours, 3 weeks, 6 weeks and 6 months postoperatively
  Total bilirubin will be used to evaluate the impacts of surgical trauma and medications on patients.
Derect bilirubin (DB) | 72 hours, 3 weeks, 6 weeks and 6 months postoperatively
  Derect bilirubin will be used to evaluate the impacts of surgical trauma and medications on patients.
Aspartate aminotransferase (AST) | 72 hours, 3 weeks, 6 weeks and 6 months postoperatively
  Aspartate aminotransferase will be used to evaluate the impacts of surgical trauma and medications on patients.
Alanine aminotransferase (ALT) | 72 hours, 3 weeks, 6 weeks and 6 months postoperatively
  Alanine aminotransferase will be used to evaluate the impacts of surgical trauma and medications on patients.
Creatinine (Cr) | 72 hours, 3 weeks, 6 weeks and 6 months postoperatively
  Creatinine will be used to evaluate the impacts of surgical trauma and medications on patients.

OTHER OUTCOMES:
Age | through study completion, an average of 6 months
  Age in years will be obtained from the electronic medical records system.
Sex | through study completion, an average of 6 months
  Sex (male or female) will be obtained from the electronic medical records system.
Operative site | through study completion, an average of 6 months
  Operative site (left or right) will be obtained from the electronic medical records system.
BMI | through study completion, an average of 6 months
  Weight (kg) and height (m) will be combined to report BMI in kg/m^2, which will be obtained from the electronic medical records system. This information will be collected by the same evaluator and used to calculate the age-corrected Charlson Comorbidity Index (aCCI), baseline ROM, HSS score and VAS score for these patients.
Time of operation | through study completion, an average of 6 months
  Inpatient data will include the operative time and time to discharge. These inpatient data will be sourced from the electronic medical records system and used to evaluate the impacts of PSIA and PLIA on the surgical process and postoperative recovery.
Operative time | through study completion, an average of 6 months
  Operative time will be sourced from the electronic medical records system and used to evaluate the impacts of PSIA and PLIA on the surgical process and postoperative recovery.
Time to discharge | through study completion, an average of 6 months
  Time to discharge will be sourced from the electronic medical records system and used to evaluate the impacts of PSIA and PLIA on the surgical process and postoperative recovery.
Incidence of Adverse events (AEs) | through study completion, an average of 6 months
  Adverse events (AEs) are adverse medical events that occur in clinical trial subjects after receiving treatment. In this study, total AEs will be mainly categorized into local AEs and systemic AEs. Local AEs include but are not limited to prolonged wound drainage (wound drainage persists on postoperative day 3, and the drainage area of the wound dressing is greater than 2×2 cm , poor wound healing and prosthetic joint infection. Systemic AEs include but are not limited to deep vein thrombosis events, systemic infection and serious adverse events such as pulmonary embolism and death.
Likert score | through study completion, an average of 6 months
  We will use a Likert scale to evaluate participants satisfaction with each treatment phase at each assessment. This scale consists of 5 levels (very dissatisfied, dissatisfied, neutral, satisfied and very satisfied) from 1 to 5. After the final follow-up, the total score on the Likert scale for each participant will represent their overall satisfaction to date. The larger the score, the more satisfactory with the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Zhang, MD, Study Director — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China